CLINICAL TRIAL: NCT02224651
Title: A Phase 1, Randomized, Double Blind, Sponsor Open, Placebo Substitution, Crossover, Single Dose Escalation Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Pf 06650833 Delivered In Multiple Formulations In Healthy Subjects Under Fasted And Fed Conditions
Brief Title: Study to Evaluate Safety and Tolerability of Single Ascending Doses of Multiple Formulations of PF-06650833 in Healthy Subjects Under Fasted and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7921001; IRAK4 FIH (Other: Alias Study Number)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- (1-1000mg) Immediate Release formulation (Experimental)
  Interventions: Drug: PF-06650833
- Immediate Release Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo
- (10-500) mg Modified Release formulation (Experimental)
  Interventions: Drug: PF-06650833
- Modified Release Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06650833 — Subjects will receive sequential single escalating doses of 1-1000 mg of Immediate Release of PF-06650833 (as solution/suspension) under fed and / or fasted conditions.
  Arms: (1-1000mg) Immediate Release formulation
Drug: Placebo — Subjects will receive sequential single escalating doses of PF-06650833 matching placebo (as solution/suspension) under fed and/ or fasted conditions.
  Arms: Immediate Release Placebo arm
Drug: PF-06650833 — Subjects will receive sequential single escalating doses of 10-500 mg of Modified Release of PF-06650833 (as capsule) under fed and / or fasted conditions.
  Arms: (10-500) mg Modified Release formulation
Drug: Placebo — Subjects will receive sequential single escalating doses of PF-06650833 matching placebo (as capsule) under fed and/ or fasted conditions.
  Arms: Modified Release Placebo arm

SUMMARY:
This single ascending dose study is the first evaluation of PF-06650833 in humans. The goals are to assess the safety, tolerability and blood levels of ascending doses of multiple formulations of PF-06650833 and to perform a preliminary assessment of the effect of food on exposure, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Screening supine blood pressure 100 mm Hg (systolic) or 50 mm Hg (diastolic); or 140 mm Hg (systolic) or 90 mm Hg (diastolic) following at least 5 minutes of supine rest. If blood pressure (BP) is 140 mm Hg (systolic) or 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
* Pulse or heart rate (HR) >100 bpm after at least 5 minutes of rest. If the pulse/HR is >100 bpm, the pulse/HR should be repeated two more times (separated by at least 2 minutes) and the average of the three pulse/HR values should be used to determine the subject's eligibility.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events and withdrawals due to treatment emergent adverse events | Baseline-5 days
Changes from baseline in vital signs ( blood pressure, pulse rate, respiratory rate and orthostatic blood pressure) | Baseline-5 days
Changes from baseline in ECG parameters (standard 12 lead ECG and telemetry) | Baseline-5 days
  Quantitative changes in ECG intervals
Incidence and magnitude of treatment emergent clinical laboratory abnormalities including hematology, chemistry (including, cardiac enzymes CK, CK MB and cardiac Troponin I), serum myoglobin, urinalysis | Baseline-5 days

SECONDARY OUTCOMES:
Cmax, Tmax, AUClast, AUCinf, CL/F, Vz/F, Cmax(dn), AUCinf(dn), AUClast(dn), t½, mean residence time (MRT) for IR and MR formulations under fasted condition | Baseline-5 days
Cmax, Tmax, AUClast, AUCinf, CL/F, Vz/F, Cmax(dn), AUCinf(dn), AUClast(dn), t½, mean residence time (MRT) for IR and MR formulations under fed condition | Baseline-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Danto SI, Shojaee N, Singh RSP, Li C, Gilbert SA, Manukyan Z, Kilty I. Safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-06650833, a selective interleukin-1 receptor-associated kinase 4 (IRAK4) inhibitor, in single and multiple ascending dose randomized phase 1 studies in healthy subjects. Arthritis Res Ther. 2019 Dec 5;21(1):269. doi: 10.1186/s13075-019-2008-6. PMID 31805989
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7921001&StudyName=Study%20to%20Evaluate%20Safety%20and%20Tolerability%20of%20Single%20Ascending%20Doses%20of%20Multiple%20Formulations%20of%20PF-06650833%20in%20Healthy%20Subjects%20Under%20Fa